CLINICAL TRIAL: NCT05542069
Title: Measurement of the Diaphragm Loading During the Training With a Inspiratory Muscle Trainer Device
Brief Title: Measurement of the Diaphragm Loading During the Training With a IMT Device
Status: Recruiting | Type: Observational
Sponsor: Clínica Basilea (Other)
Responsible Party: Principal Investigator, Dario Villalba, clinical professor, Clínica Basilea
Other Study IDs: Basilea00000000000000001
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Threshold IMT (Inspiratory muscle trainer) by Philips — Apply a resistive load with the IMT device according the maximal inspiratory pressure of each subject.

SUMMARY:
It is well known that the the training with the IMT device increases the Maximal Inspiratory Pressure. Nonetheless, there are doubts about which muscles are involved during this training. The aim of this study is to determine the diaphragm loading of healthy subjects during the training with a IMT device from a low . Therefore, each subject will be monitored using esophageal and gastric manometry.

DETAILED DESCRIPTION:
This study has a quasi-experimental design. The investigators will recruit ten healthy adult volunteers without anticoagulation or esophageal lesions, after signing a consent form.

After checking the appropriate correct position of each catheter, each subject will use the IMT device throughout different randomized loads (percentages of the maximal inspiratory pressure, counting by tens from 10% to 100%). FluxMed® GrT MBMed respiratory mechanic monitor will be used. Each percentage of resistive load will be maintained for 5 inspirations. Meanwhile, an operator will register the esophageal pressure,the gastric pressure and the transdiaphragmatic pressure. Diaphragm collaboration in each percentage of resistive load will be determine by calculating the relation between the gastric pressure and the transdiaphragmatic pressure (∆Pgas/∆Pdi).

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* healthy subjects

Exclusion Criteria:

* without anticoagulation
* without esophageal lesions
* without airway lesions
* without spirometry alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Diaphragm intervention during a certain percentage of resistive load with a IMT device | 1 year
  The diaphragm intervention is determined by the relation of the gastric pressure and the transdiaphragmatic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Dario Villalba, PT, Study Director — Clinica Basilea
Locations (1):
- Clinica Basilea, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No